CLINICAL TRIAL: NCT03404167
Title: A Phase 1 Clinical Trial to Evaluate the Plasma Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of Zoliflodacin in Healthy Male and Female Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability and Plasma PK of a Single Oral Dose of Zoliflodacin in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0118; HHSN272201500005I
Record Dates: First submitted 2018-01-04; First posted 2018-01-19 (Actual); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-01-11

CONDITIONS: Gonorrhoea
Keywords: ETX0914; Plasma Pharmacokinetic; Safety; Tolerability; Zoliflodacin
MeSH Terms: conditions — Gonorrhea | interventions — zoliflodacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zoliflodacin (Experimental): 4 g (2 sachets of 2 g) of zoliflodacin orally in the morning of Day 1 after 8 hours of fasting, n=8
  Interventions: Drug: AZD0914

INTERVENTIONS:
Drug: AZD0914 — Zoliflodacin (also known as AZD0914 and ETX0914), is a spiropyrimidinetrione antibacterial agent

SUMMARY:
The trial is to evaluate the pharmacokinetics and safety profiles of the single-dose of zoliflodacin in eight healthy male or female subjects ages 18 to 45 years inclusive. All subjects will be dosed in the morning of Day 1 in a staggered fashion with a minimum of several minutes apart. Each subject will receive a single 4g dose of zoliflodacin (2 x 2 g sachets of zoliflodacin) after at least an 8-h fast, which will continue for at least 4 h after dosing. Consumption of water will be permitted during the fasting period. Subjects will be monitored as inpatients in the Clinical Trial Unit (CTU) up to Day 4 and at the Final Visit (Day 8 ± 2). Study duration is approximately 4 weeks with subject participation duration up to 10 days (from dosing to final visit). The primary objective of this study is to evaluate the plasma PK of zoliflodacin after administration of a single 4-g oral dose under fasting conditions.

DETAILED DESCRIPTION:
The trial will be performed as an open-label, non-randomized, single-dose design in eight healthy male or female subjects ages 18 to 45 years inclusive to evaluate the pharmacokinetics and safety profiles of the zoliflodacin formulation. All subjects will be dosed in the morning of Day 1 in a staggered fashion with a minimum of several minutes apart. Each subject will receive a single 4g dose of zoliflodacin (2 x 2 g sachets of zoliflodacin) after at least an 8-h fast, which will continue for at least 4 h after dosing. Consumption of water will be permitted during the fasting period. Subjects will be monitored as inpatients in the Clinical Trial Unit (CTU) up to Day 4 and at the Final Visit (Day 8 ± 2). Study duration is approximately 4 weeks with subject participation duration up to 10 days (from dosing to final visit). The primary objective of this study is to evaluate the plasma PK of zoliflodacin after administration of a single 4-g oral dose under fasting conditions. The secondary objective is to evaluate the safety and tolerability of a single 4-g oral dose of zoliflodacin.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form (ICF) understood and signed before initiating any study procedures
2. Healthy male or female, as assessed by the authorized site clinician (listed on FDA Form 1572)
3. Willingness to comply with and be available for all protocol procedures including inpatient confinement for about 4 days and availability for follow-up for the duration of the trial
4. Aged 18 to 45 years inclusive on the day of study drug dosing
5. Body Mass Index (BMI) > / = 18.5 and < / = 30 kg/m^2 and weight > / = 50 kg (110 lbs.) and < / = 100 kg (220 lbs.)
6. In female subjects of childbearing potential, a negative serum pregnancy test at Screening Visit and on Day -1

   - Note: A woman is considered of childbearing potential unless post-menopausal (> / = 1 year without menses without other known or suspected cause and with a FSH level in the menopausal range), or surgically sterilized (hysterectomy, salpingectomy, oophorectomy or tubal ligation/occlusion)
7. If female, not pregnant, not breast feeding, and not planning on becoming pregnant during the trial and for 30 days after study participation
8. Females of childbearing potential and males agree to use acceptable contraception for the duration of the trial and for 30 days (females) or 90 days (males) after final study visit

   - Note: A highly effective method of birth control is defined as one with a low failure rate (i.e., less than 1 percent per year) according to the CDC criteria. These include progestin implants, intrauterine devices (IUDs), surgical (hysterectomy, salpingectomy, oophorectomy or tubal ligation/occlusion; vasectomy), or abstinence. Use of methods with higher failure rate (such as progestin injectables, combined oral hormonal contraceptives, condoms, and diaphragms) will not be acceptable when used alone, but they could be considered if used in combination with another method (e.g., a female using combined oral contraceptives if her male partner is sterile, or if she and her non-sterile male partner use a double-barrier method), after consultation with the DMID Medical Officer
9. Male subjects must agree to refrain from sperm donation for the duration of the trial and for 90 days after Final Visit
10. Laboratory tests are in the normal reference range with acceptable exceptions
11. Vital signs are within the acceptable range
12. Has adequate venous access for blood collection
13. Urine drug screen is negative for tested substances
14. Alcohol test (breathalyzer) is negative
15. Willing to abstain from alcohol consumption for 2 days before Day -1 and during the trial

Exclusion Criteria:

1) History of a chronic medical or surgical condition that would interfere with the accurate assessment of the trial's objectives or increase the subject's risk profile

* Note: Chronic medical conditions include: diabetes mellitus; asthma requiring use of medication in the year before screening; autoimmune disorder such as lupus erythematosus, Wegener's, rheumatoid arthritis, thyroid disease; cardiovascular disease, including coronary artery disease or cerebrovascular disease, or surgery; syncope related to cardiac arrhythmia or unexplained; chronic hypertension; malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease, myopathy, or neuropathy; gastrointestinal or biliary surgery.

  2) History of hypersensitivity or severe allergic reaction of any type to medications, bee stings, food, or environmental factors
* Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema 3) Active allergic symptoms to seasonal and animal allergens that require treatment 4) A marked baseline prolongation of ECG intervals, or HR < 45 bpm or > 100 bpm on ECG measurements
* Note: The following are considered prolonged ECG intervals: QTc/QTcF > 449 msec in males and females; PR > 209 msec; and QRS > 110 msec 5) Clinically significant abnormal ECG results
* Note: Clinically significant abnormal ECG results include: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained atrial or ventricular arrhythmia; two premature ventricular contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; evidence of a previous myocardial infarction (MI), left ventricular hypertrophy (LVH), or more than minor non-specific ST-T wave changes; or any condition deemed clinically significant by a study investigator 6) Abnormal renal function
* Note: Normal renal function is defined as normal creatinine and normal estimated glomerular filtration rate (eGFR) [i.e., > 80.0 mL/min] values according to Cockroft-Gault 7) Positive serology results for HIV, HBsAg, or HCV 8) Febrile illness with temperature > 37.6°C for < 7 days before dosing 9) Donated whole blood or blood products within 60 days before dosing, or plans to donate before Final Visit (Day 8 ± 2)
* Note: Blood products include RBCs, WBCs, platelets, and plasma 10) Known allergic reactions to any of the study drug components present in the formulation or in its processing, as listed in the IB 11) Treatment with another investigational product within 30 days of dosing or 5 half-lives or twice the duration of the biological effect of the study drug (whichever is longer)
* Note: Investigational products include a drug, vaccine, biologic, device or blood product 12) Active drug or alcohol use, abuse, or dependence within 12 months before Screening Visit that, in the opinion of the investigator, would interfere with adherence to study requirements 13) Use of any prescription medication within 30 days before dosing or planned use during the study period except as noted below and approved by the designated study clinician
* Note 1: Prohibited medications include moderate or strong CYP3A4 inducers; antibiotics; injectable or oral antidiabetic drugs; anti-lipid drugs; immunosuppressive agents; immune modulators; oral corticosteroids; anti-neoplastic agents; any vaccine (licensed or investigational) except licensed influenza vaccine during the flu season, which is allowed 7 days before or after dosing
* Note 2: Allowed medications include: oral contraceptives; H1 antihistamines; topical/ intranasal corticosteroids; nonsteroidal anti-inflammatory drugs [NSAIDS]; licensed influenza vaccine during the flu season, 7 days before or after dosing.

  14) Use of any non-prescription medication, herbal preparation, or nutritional supplement within 15 days before dosing or planned use during the study unless approved by the study clinician
* Note: Exceptions: St. John's wart is not allowed within 30 days of dosing, vitamins and OTC medications taken for a brief period (<48 h) for the treatment of common symptoms (such as headache, indigestion, muscle pain) may be allowed as approved by the designated study clinician 15) Intake of caffeinated beverages or food within 72 h before dosing or a history of high caffeine consumption (e.g., in the last 4 months drinking > 5 cups of coffee/day) 16) Smoking or use of tobacco or nicotine-containing products within 15 days before dosing 17) Engagement in strenuous exercise within 15 days before dosing (e.g., marathon running, long distance cycling, weight lifting) and during the study period 18) Any specific behavioral or clinical condition that in the judgment of the investigator precludes participation because it could affect compliance with study procedures or subject safety 19) Plans to enroll or is already enrolled in another clinical trial that could interfere with safety assessment of the study drug at any time during the study period
* Note: Includes trials that have a study intervention such as a drug, biologic, or device 20) Is a study site employee or staff member who is paid entirely or partially by the OCRR/NIAID contract for the DMID-funded trial
* Note: Site employees or staff include the PIs, sub-investigators, or staff who are supervised by the PI or sub-investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services - Overland Park, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed at a commercial phase 1 unit. Recruitment opened on February 2, 2018 and all eight participants were consented and screened for meeting eligibility criteria prior to enrollment and dosing on Feb 23, 2018.
Pre-assignment Details: This was an open-label, non-randomized single-dose oral treatment of eligible participants followed by follow up to eight days after dosing.
Groups:
- Zoliflodacin: 4 g (2 sachets of 2 g) of zoliflodacin orally in the morning of Day 1 after 8 hours of fasting
  AZD0914: Zoliflodacin (also known as AZD0914 and ETX0914), is a spiropyrimidinetrione antibacterial agent
Period: Overall Study
Arm/Group | Zoliflodacin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants are included in the baseline analysis population.
Groups:
- Zoliflodacin: 4 g (2 sachets of 2 g) of zoliflodacin administered orally to eight participants in the morning of Day 1 after 8 hours of fasting
  AZD0914: Zoliflodacin (also known as AZD0914 and ETX0914), is a spiropyrimidinetrione antibacterial agent
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.50 (1.59)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Zoliflodacin
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
ng/mL | 20863 (7129)

2. Primary Outcome: Time of Maximum Observed Concentration (Tmax) of Zoliflodacin
Description: Tmax was defined as the time at which the maximum concentration (Cmax) occurs in plasma computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
hour | 4 (3)

3. Primary Outcome: Area Under the Concentration Time-curve From Time Zero to Infinity (AUC(0-infinity)) for Zoliflodacin
Description: AUC(0-8) was defined as the total area under the concentration-time curve from dosing (time 0) taken to the limit as the end time becomes arbitrarily large. AUC(0-8) and was calculated by adding AUC(0-last) to an extrapolated value equal to the last measured concentration greater than the lower limit of quantification of the bioanalytical assay divided by the terminal phase elimination rate constant (Ke) computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: h x ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
h x ng/mL | 226750 (85336)

4. Primary Outcome: Area Under the Concentration Time-curve From Time Zero to the Last Concentration Above the Lower Limit of Quantitation (AUC(0-last)) for Zoliflodacin
Description: AUC(0-last) was defined as the area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: h x ng/mL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
h x ng/mL | 226500 (85340)

5. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Zoliflodacin
Description: Apparent volume of distribution during terminal phase (Vz/F) after non-intravenous administration was calculated as (CL/F)/ Ke computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Liter | 183.6 (58.8)

6. Primary Outcome: Apparent Oral Clearance (CL/F) of Zoliflodacin
Description: Apparent oral clearance (CL/F) computed as Dose/Area under the curve (AUC) from time zero to infinity (0-8) computed from concentrations that were measured using a validated high-performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) method.
Time Frame: Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
L/h | 19.9 (7.0)

7. Primary Outcome: Elimination Rate Constant (Ke) of Zoliflodacin
Description: The terminal phase elimination rate constant (Ke) was defined as the first-order rate constant describing the rate of decrease of drug concentration in the terminal phase (defined as the terminal region of the PK curve where drug concentration follows first-order elimination kinetics) computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
1/hour | 0.108 (0.011)

8. Primary Outcome: Terminal Elimination Half-life (t1/2) of Zoliflodacin
Description: The apparent terminal elimination half-life (t1/2) was defined as the time required for the drug concentration to decrease by a factor of one-half in the terminal phase computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: From Day 1 to Day 4
Population: The analysis population consists of all eight participants.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
hour | 6.5 (0.6)

9. Secondary Outcome: Changes From Baseline for White Blood Cells With Differentials and Platelets
Description: Change from baseline calculated by subtracting the Day -1 (baseline) hematology measurement from the Day 4 hematology measurement. Hematology parameters included white blood cell count, differential (absolute counts of neutrophils, lymphocytes, monocytes, eosinophils, and basophils), and platelet count.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
10^9/L
  Leukocytes | -0.659 (1.668)
  Neutrophils | -0.118 (0.950)
  Lymphocytes | -0.465 (0.689)
  Monocytes | -0.036 (0.075)
  Eosinophils | -0.035 (0.096)
  Basophils | -0.008 (0.019)
  Platelets | -7.1 (21.9)

10. Secondary Outcome: Changes From Baseline Hematocrit
Description: Change from baseline calculated by subtracting the Day -1 (baseline) hematocrit measurement from the Day 4 hematocrit measurement.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
percentage | 1.36 (1.68)

11. Secondary Outcome: Changes From Baseline Hemoglobin
Description: Change from baseline calculated by subtracting the Day -1 (baseline) hemoglobin measurement from the Day 4 hemoglobin measurement.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
g/dL | 0.46 (0.66)

12. Secondary Outcome: Changes From Baseline Red Blood Cell Count
Description: Change from baseline calculated by subtracting the Day -1 (baseline) red blood cell count measurement from the Day 4 red blood cell count measurement.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
10^12/L | 0.150 (0.201)

13. Secondary Outcome: Changes From Baseline for Albumin and Total Protein
Description: Change from baseline calculated by subtracting the Day -1 (baseline) albumin or total protein measurement from the Day 4 albumin or total protein measurement.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
g/dL
  Albumin | 0.02 (0.23)
  Total Protein | 0.11 (0.29)

14. Secondary Outcome: Change From Baseline for Alkaline Phosphatase (AP), Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST)
Description: Change from baseline calculated by subtracting the Day -1 (baseline) AP, ALT, or AST measurement from the Day 4 AP, ALT, or AST measurement.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
U/L
  Alkaline Phosphatase | -3.1 (7.2)
  Alanine Aminotransferase | 1.5 (4.3)
  Aspartate Aminotransferase | -0.8 (2.7)

15. Secondary Outcome: Change From Baseline for Blood Urea Nitrogen (BUN), Serum Creatinine, Glucose (Fasting at Least 4h), Magnesium, Total and Direct Bilirubin
Description: Change from baseline calculated by subtracting the Day -1 (baseline) serum chemistry measurement from the Day 4 serum chemistry measurement. Serum chemistry tests for this outcome measure included BUN, creatinine, fasting glucose, magnesium, total bilirubin, and direct bilirubin.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Days -1 and 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
mg/dL
  BUN | -3.0 (2.1)
  Creatinine | 0.05 (0.08)
  Glucose (fasting) | -2.6 (3.2)
  Magnesium | -0.01 (0.08)
  Total Bilirubin | 0.03 (0.31)
  Direct Bilirubin | -0.01 (0.06)

16. Secondary Outcome: Changes From Baseline for Sodium, Potassium, Chloride and Bicarbonate
Description: Change from baseline calculated by subtracting the Day -1 (baseline) serum chemistry measurement from the Day 4 serum chemistry measurement. Serum chemistry tests for this outcome measure included sodium, potassium, chloride, and bicarbonate.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had safety labs collected on Day -1 and Day 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
mmol/L
  Sodium | -1.1 (1.7)
  Potassium | -0.24 (0.36)
  Chloride | -3.6 (0.9)
  Bicarbonate | 0.5 (1.2)

17. Secondary Outcome: Changes From Baseline for Blood Pressure - Systolic
Description: Change from baseline in systolic blood pressure calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, and 4 h after dosing, and on Day 2, Day 3, Day 4, and Day 8. Vital signs were measured after supine for at least 10 minutes.
Time Frame: From Day -1 through Day 8
Population: Any participants who received study product and had vital signs collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
mmHg
  1 Hour | 1.1 (3.9)
  2 Hour | 0 (5.9)
  4 Hour | -3.9 (6.0)
  Day 2 | -1.1 (5.6)
  Day 3 | -3.6 (7.4)
  Day 4 | 0.5 (6.5)
  Day 8 | 2.4 (11.4)

18. Secondary Outcome: Changes From Baseline for Blood Pressure - Diastolic
Description: Change from baseline in diastolic blood pressure calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, and 4 h after dosing, and on Day 2, Day 3, Day 4, and Day 8. Vital signs were measured after supine for at least 10 minutes.
Time Frame: From Day -1 through Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
mmHg
  1 Hour | 0.1 (5.5)
  2 Hour | -5.3 (6.1)
  4 Hour | -4.5 (6.3)
  Day 2 | -2.8 (7.5)
  Day 3 | -4.1 (6.5)
  Day 4 | 0.0 (6.3)
  Day 8 | -1.0 (10.7)

19. Secondary Outcome: Changes From Baseline in Oral Temperature
Description: Change from baseline in temperature calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, and 4 h after dosing, and on Day 2, Day 3, Day 4, and Day 8. Vital signs were measured after supine for at least 10 minutes.
Time Frame: From Day -1 through Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degress C
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Degress C
  1 Hour | -0.04 (0.29)
  2 Hour | 0.03 (0.17)
  4 Hour | 0.01 (0.24)
  Day 2 | -0.06 (0.17)
  Day 3 | -0.09 (0.16)
  Day 4 | 0.06 (0.21)
  Day 8 | -0.04 (0.23)

20. Secondary Outcome: Changes From Baseline in Pulse Rate
Description: Change from baseline in pulse rate calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, and 4 h after dosing, and on Day 2, Day 3, Day 4, and Day 8. Vital signs were measured after supine for at least 10 minutes.
Time Frame: From Day -1 through Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Beats per minute
  1 Hour | -3.8 (11.7)
  2 Hour | -0.4 (14.0)
  4 Hour | -3.5 (12.6)
  Day 2 | -4.3 (12.8)
  Day 3 | -1.8 (8.7)
  Day 4 | -1.9 (13.3)
  Day 8 | 1.9 (14.0)

21. Secondary Outcome: Changes From Baseline for Respiratory Rate
Description: Change from baseline in respiratory rate calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, and 4 h after dosing, and on Day 2, Day 3, Day 4, and Day 8. Vital signs were measured after supine for at least 10 minutes.
Time Frame: From Day -1 through Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Breaths per minute
  1 Hour | 0.3 (1.7)
  2 Hour | 1.0 (2.1)
  4 Hour | 0.8 (2.4)
  Day 2 | 0.8 (1.0)
  Day 3 | 0.5 (0.9)
  Day 4 | 0.5 (1.4)
  Day 8 | 0.5 (1.8)

22. Secondary Outcome: Changes From Baseline in ECG: PR Interval (Interval From Onset of P-wave to the Onset of the QRS Complex)
Description: Change from baseline in ECG PR Interval calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, and 72 h after dosing.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had an ECG collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
msec
  1 Hour | 4.0 (8.6)
  2 Hour | 2.3 (6.6)
  4 Hour | 1.5 (7.9)
  72 Hour | 6.9 (7.7)

23. Secondary Outcome: Changes From Baseline in ECG: QRS Duration (Time From the Start of the Q-wave to the End of the S-wave)
Description: Change from baseline in ECG QRS Duration calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, and 72 h after dosing.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had an ECG collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
msec
  1 Hour | -0.3 (3.3)
  2 Hour | 0.5 (2.7)
  4 Hour | -0.1 (2.7)
  72 Hour | 1.0 (3.9)

24. Secondary Outcome: Changes From Baseline in ECG: QTcF Interval (QT Interval Corrected by Fridericia's Formula)
Description: Change from baseline in ECG QTcF Interval calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, and 72 h after dosing.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had an ECG collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
msec
  1 Hour | 1.8 (13.6)
  2 Hour | 6.8 (13.2)
  4 Hour | 4.0 (11.6)
  72 Hour | -2.6 (11.2)

25. Secondary Outcome: Changes From Baseline in ECG: QT Interval (Interval From Onset of the Q-wave to the End of the T-wave)
Description: Change from baseline in ECG QT Interval calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, and 72 h after dosing.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had an ECG collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
msec
  1 Hour | -1.1 (13.8)
  2 Hour | 4.6 (15.6)
  4 Hour | 3.6 (10.8)
  72 Hour | -6.3 (8.8)

26. Secondary Outcome: Changes From Baseline in ECG: RR Interval (Interval From the Peak of the R Wave of a QRS Complex to the Peak of the R Wave of the Next QRS Complex)
Description: Change from baseline in ECG RR Interval calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, and 72 h after dosing.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had an ECG collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
msec
  1 Hour | -23.3 (120.9)
  2 Hour | -20.3 (122.3)
  4 Hour | -7.0 (64.5)
  72 Hour | -30.1 (77.3)

27. Secondary Outcome: Changes From Baseline in ECG: Ventricular Rate
Description: Change from baseline in ECG Ventricular Rate calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, and 72 h after dosing.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had an ECG collected on Day -1 and at least one time point post dose.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
beats per minute
  1 Hour | 1.4 (8.0)
  2 Hour | 0.9 (6.4)
  4 Hour | 0.0 (3.6)
  72 Hour | 1.8 (4.9)

28. Secondary Outcome: Changes From Baseline for Occult Blood Via Dipstick
Description: Urine for the clinical laboratory test was collected on Day -1 and Day 4. The results for occult blood were reported in categorical results. The possibilities were negative, trace, 1+, 2+, and 3+.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had urine collected on Day -1 and Day 4.
Measure: Number; unit: participants
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
participants | 0

29. Secondary Outcome: Changes From Baseline for Glucose Via Dipstick
Description: Urine for the clinical laboratory test was collected on Day -1 and Day 4. The results for glucose were reported in categorical results. The possibilities were negative, trace, 1+, 2+, and 3+.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had urine collected on Day -1 and Day 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Participants | 0

30. Secondary Outcome: Changes From Baseline for Protein Via Dipstick
Description: Urine for the clinical laboratory test was collected on Day -1 and Day 4. The results for protein were reported in categorical results. The possibilities were negative, trace, 1+, 2+, and 3+.
Time Frame: From Day -1 through Day 4
Population: Any participants who received study product and had urine collected on Day -1 and Day 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Participants | 0

31. Secondary Outcome: Occurrence of Unsolicited Treatment-emergent Adverse Events
Description: Adverse events are defined as any untoward medical occurrence regardless of its causal relationship to the study treatment.
Time Frame: From study product administration (Day 1) to Day 8
Population: Any participants who received study product
Measure: Count of Participants; unit: Participants
Groups:
- Zoliflodacin: 4 g (2 sachets of 2 g) of zoliflodacin administered orally to eight participants in the morning of Day 1 after 8 hours of fasting.
  AZD0914: Zoliflodacin (also known as AZD0914 and ETX0914), is a spiropyrimidinetrione antibacterial agent
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Participants | 8

32. Secondary Outcome: Occurrence of Treatment-emergent Serious Adverse Events
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect.
Time Frame: From study product administration (Day 1) to Day 8
Population: Any participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoliflodacin
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: Unsolicited Adverse Events and serious adverse events (SAEs) were collected from study product administration to Day 8.
Description: Treatment emergent adverse events were defined as new events post-dose, or worsening of existing conditions post-dose. The adverse events were captured by changes in laboratory values, vital signs, ECGs and unsolicited adverse events immediately post dose to Day 8 or early termination whichever came first.
Arm/Group | Zoliflodacin
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoliflodacin (N=8)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 6 (6)
HEART RATE DECREASED (Investigations) | 4 (4)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03404167/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT03404167/SAP_001.pdf